CLINICAL TRIAL: NCT00000845
Title: A Phase I Safety and Immunogenicity Trial of UBI HIV Lipopeptide Vaccine Component P3C541b in HIV-1 Seronegative Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 021
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: P3C541b Lipopeptide

SUMMARY:
To evaluate an HIV synthetic lipopeptide candidate vaccine component, P3C541b, at two dose levels, administered subcutaneously (s.c.) in a randomized, double-blind, placebo controlled study.

DETAILED DESCRIPTION:
The prospective volunteers will be screened and HLA typed for Class I MHC haplotypes. Only volunteers possessing HLA alleles A33, B8, B27, B35 or Bw62 or any combination thereof will be enrolled in the study. Subjects will be allocated to 1 of 2 study groups. Group 1 will receive 70 mcg of P3C541b or the placebo and Group II will receive 350 mcg of P3C541b or the placebo. NOTE: Enrollment for Group II wil not begin until at least 5 Group I participants have reached day 14 without serious adverse events.

ELIGIBILITY:
Inclusion Criteria

Patients must have or be:

* Healthy
* Negative ELISA for HIV.
* One or more HLA alleles:
* A33, B8, B27, B35, or Bw62.
* Negative for Hepatitis B surface antigen.
* Normal urine dipstick.
* Normal history and physical examination.
* Availability for follow-up planned duration of the study (12 months).
* Viable EBV line prior to enrollment.

Risk behavior: Required:

* Lower risk sexual behavior as defined by AVEG.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Medical or psychiatric condition or occupational responsibilities, which preclude subject compliance with the protocol (e.g., recent suicidal ideation or present psychosis).
* Active syphilis. NOTE: If the serology is documented to be false positive due to a remote (> 6 months) treated infection, the volunteer is eligible.
* Hepatitis B surface antigenemia.
* Active tuberculosis. NOTE: Volunteers with a positive PPD and a normal chest X-Ray showing no evidence of TB and not requiring INH therapy are eligible.

Patients with any of the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, malignancy, autoimmune disease.
* History of cancer, unless there has been surgical excision followed by a sufficient observation period to give a reasonable assurance of a cure.
* History of anaphylaxis or history of other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance, requiring hospitalization or emergent medical care.
* History of suicide attempts or past psychosis.

Prior Medication:

Excluded:

* History of use of immunosuppressive medication.
* Live attenuated vaccines within 60 days of study.

NOTE:

* Medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal) are not exclusionary but should be given at least 2 weeks away from HIV immunizations.
* Use of experimental agents within 30 days prior to study.

Prior Treatment:

Excluded:

* Receipt of blood products or immunoglobulin in the past 6 months.

Risk Behavior:

Excluded:

* Subjects with identifiable higher risk behavior for HIV infection as determined by screening questionnaire designed to identify risk factors for HIV infection.
* History of injection drug use within the last 12 months prior to enrollment.
* Higher or intermediate risk sexual behavior as defined by AVEG.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Schwartz D, Study Chair
Locations (3):
- United States (3):
  - Johns Hopkins Univ / School of Hygiene & Public Health, Baltimore, Maryland
  - Vanderbilt Univ Hosp, Nashville, Tennessee
  - Univ of Washington / Pacific Med Ctr, Seattle, Washington